CLINICAL TRIAL: NCT06637072
Title: A Phase 4, Open-Label, Single-Group, Multicenter Study in Adult Participants With Chronic Inflammatory Demyelinating Polyneuropathy Who Transition From Treatment With Intravenous Immunoglobulin to Efgartigimod PH20 SC
Brief Title: A Study to Assess Adults With CIDP Transitioning From IVIg to Efgartigimod PH20 SC
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARGX-113-2406
Record Dates: First submitted 2024-10-07; First posted 2024-10-15 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Efgartigimod PH20 SC (Experimental): Participants start efgartigimod PH20 SC treatment after discontinuing IVIg
  Interventions: Biological: Efgartigimod PH20 SC

INTERVENTIONS:
Biological: Efgartigimod PH20 SC — Subcutaneous injection of efgartigimod PH20 SC

SUMMARY:
This study will measure how adults with CIDP receiving IVIg treatment adjust to efgartigimod PH20 SC. The study duration for each participant will be approximately 17 to 19 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age and the local legal age of consent
* Is diagnosed with CIDP (confirmed or possible CIDP) according to the criteria of the European Academy of Neurology/Peripheral Nerve Society
* Is being treated with IVIg every 3-6 weeks, on a stable dose and dosing interval (between 0.5-2 g/kg) for at least 3 doses
* If receiving oral corticosteroids, this should be at a stable dose of less than 20 mg a day or less than 40 mg every other day, for at least a month.
* If receiving nonsteroidal immunosuppressive medication, this should be at a stable dose for at least 3 months

Exclusion Criteria:

* Besides the indication under study, known autoimmune disease or any medical condition that would interfere with an accurate assessment of clinical symptoms of CIDP or puts the participant at undue risk
* Types of other polyneuropathy other than CIDP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-02-23 (Estimated); Study Completion 2026-02-23 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who begin treatment with efgartigimod PH20 SC within 1 week after stopping IVIg therapy and are still receiving efgartigimod PH20 SC at the end of the 12-week treatment period | Up to 12 weeks

SECONDARY OUTCOMES:
Changes from baseline in EQ-5D-5L scores over time | Up to 12 weeks
Changes from baseline in TSQM-9 scores over time | Up to 12 weeks
Changes from baseline in PGI-C scores over time | Up to 12 weeks
Changes from baseline in PGI-S scores over time | Up to 12 weeks
Incidence of (S)AEs | Up to 16 weeks

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Neurology Associates PA, Maitland, Florida
  - Visionary Investigators Network, Miami, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Velocity Clinical Research, Lafayette, Louisiana
  - SRI International - ClinEdge, Plymouth, Michigan
  - Velocity Clinical Research, Raleigh, North Carolina
  - Erlanger Neuroscience Institute, Chattanooga, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - National Neuromuscular Research Institute, Austin, Texas
  - Horizon Clinical Research: Gill Neuroscience, Cypress, Texas
  - Northwest Houston Neurology - Cypress, Cypress, Texas
  - Cedar Health Research - Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No